CLINICAL TRIAL: NCT06362850
Title: Tele-Support for Emergency Medical Technicians Dealing with Pediatric Cardiac Arrest: a Randomized, Simulation-based Study
Brief Title: Tele-Support for Emergency Medical Technicians
Acronym: POHCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Ludwig Boltzmann Institute Digital Health and Patient Safety (Other)
Responsible Party: Principal Investigator, Christina Hafner, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1253/2023
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrest
Keywords: simulation; pediatric out-of-hospital cardiac arrest; advanced life support; eye tracking; cognitive load; emergency medicine; patient safety; telemedicine; anaesthesiology
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: In a manikin-based simulation study, the participants will be randomized to either performing the scenario with tele-support or without tele-support (80 participants 40 groups, 20 groups with tele-support, 20 groups without tele-support).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No-Support (No Intervention): Participants randomized to Group 1 will perform the simulation scenario without tele-support.
- Tele-Support (Other): Participants randomized to Group 2 will perform the simulation scenario with tele-support.
  Interventions: Other: Tele-support

INTERVENTIONS:
Other: Tele-support — via real-time audio-video connection through an experienced physician
  Arms: Tele-Support

SUMMARY:
In this manikin-based simulation study the impact of tele-support during a simulated pediatric out-of-hospital cardiac arrest scenario on emergency medical technicians' guideline adherence, on gaze behavior as well as on performance of resuscitation management and cognitive load will be analyzed.

DETAILED DESCRIPTION:
80 emergency medical technicians (EMT) will take part in this simulation study. The participants will be confronted with a scenario of an 8-year old boy, while wearing eye tracking glasses. In a parallel group design, the teams will be randomly assigned to a group performing advanced life support (ALS) without further support (group 1) or with additional tele-support (group 2). In case of support, an emergency physician assists the team performing the cardiopulmonary resuscitation management via a real-time remote connection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Active work as an emergency medical technician

Exclusion Criteria:

* Pregnancy
* Prior knowledge of study setting or simulation scenario

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
guideline adherence | Day 1
  checklist (scale of 0-15 points)

SECONDARY OUTCOMES:
gaze behavior | Day 1
  dwell time in predefined areas of interest and fixation count
teamwork performance | Day 1
  Team Emergency Assessment Measure (11 items on scale 0-4 for components leadership, team work and task management resulting in a total score with scale 0-44; scale 1-10 for overall global rating)
cognitive load | Day 1
  NASA Taskload Index (scale of 0-20 points)
Performance of cardiopulmonary resuscitation | Day 1
  Chest compressions (time to 1st compression, depth, frequency, total hands-off period); defibrillator: time to 1st rhythm analysis; ventilation: time to 1st ventilation, airway management; intravenous access: time to drug application; reversible causes: time to discussing potential reversible causes for cardiac arrest
Technical feasibility | Day 1
  time of detection of visual attention through eye-tracking glasses
Usability | Day 1
  Questionnaire (5-point Likert scale) on usability of tele-support and eye-tracking glasses

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hafner, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Anesthesia, General Intensive Care and Pain Management,Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available to other researchers.

REFERENCES:
- [Background] Drummond D, Arnaud C, Guedj R, Duguet A, de Suremain N, Petit A. Google Glass for Residents Dealing With Pediatric Cardiopulmonary Arrest: A Randomized, Controlled, Simulation-Based Study. Pediatr Crit Care Med. 2017 Feb;18(2):120-127. doi: 10.1097/PCC.0000000000000977. PMID 28165347
- [Background] Reis AG, Nadkarni V, Perondi MB, Grisi S, Berg RA. A prospective investigation into the epidemiology of in-hospital pediatric cardiopulmonary resuscitation using the international Utstein reporting style. Pediatrics. 2002 Feb;109(2):200-9. doi: 10.1542/peds.109.2.200. PMID 11826196
- [Background] Gupta P, Tang X, Gall CM, Lauer C, Rice TB, Wetzel RC. Epidemiology and outcomes of in-hospital cardiac arrest in critically ill children across hospitals of varied center volume: a multi-center analysis. Resuscitation. 2014 Nov;85(11):1473-9. doi: 10.1016/j.resuscitation.2014.07.016. Epub 2014 Aug 7. PMID 25110249
- [Background] Knudson JD, Neish SR, Cabrera AG, Lowry AW, Shamszad P, Morales DL, Graves DE, Williams EA, Rossano JW. Prevalence and outcomes of pediatric in-hospital cardiopulmonary resuscitation in the United States: an analysis of the Kids' Inpatient Database*. Crit Care Med. 2012 Nov;40(11):2940-4. doi: 10.1097/CCM.0b013e31825feb3f. PMID 22932398
- [Background] Cheng A, Nadkarni VM, Mancini MB, Hunt EA, Sinz EH, Merchant RM, Donoghue A, Duff JP, Eppich W, Auerbach M, Bigham BL, Blewer AL, Chan PS, Bhanji F; American Heart Association Education Science Investigators; and on behalf of the American Heart Association Education Science and Programs Committee, Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Cardiovascular and Stroke Nursing; and Council on Quality of Care and Outcomes Research. Resuscitation Education Science: Educational Strategies to Improve Outcomes From Cardiac Arrest: A Scientific Statement From the American Heart Association. Circulation. 2018 Aug 7;138(6):e82-e122. doi: 10.1161/CIR.0000000000000583. PMID 29930020
- [Background] Scheans P. Telemedicine for neonatal resuscitation. Neonatal Netw. 2014 Sep-Oct;33(5):283-7. doi: 10.1891/0730-0832.33.5.283. PMID 25161137
- [Background] Agarwal AK, Gaieski DF, Perman SM, Leary M, Delfin G, Abella BS, Carr BG. Telemedicine REsuscitation and Arrest Trial (TREAT): A feasibility study of real-time provider-to-provider telemedicine for the care of critically ill patients. Heliyon. 2016 Apr 20;2(4):e00099. doi: 10.1016/j.heliyon.2016.e00099. eCollection 2016 Apr. PMID 27441272
- [Background] Berrens ZJ, Gosdin CH, Brady PW, Tegtmeyer K. Efficacy and Safety of Pediatric Critical Care Physician Telemedicine Involvement in Rapid Response Team and Code Response in a Satellite Facility. Pediatr Crit Care Med. 2019 Feb;20(2):172-177. doi: 10.1097/PCC.0000000000001796. PMID 30395026
- [Background] Siebert JN, Ehrler F, Combescure C, Lovis C, Haddad K, Hugon F, Luterbacher F, Lacroix L, Gervaix A, Manzano S; PedAMINES Trial Group. A mobile device application to reduce medication errors and time to drug delivery during simulated paediatric cardiopulmonary resuscitation: a multicentre, randomised, controlled, crossover trial. Lancet Child Adolesc Health. 2019 May;3(5):303-311. doi: 10.1016/S2352-4642(19)30003-3. Epub 2019 Feb 21. PMID 30797722
- [Background] Siebert JN, Lacroix L, Cantais A, Manzano S, Ehrler F. The Impact of a Tablet App on Adherence to American Heart Association Guidelines During Simulated Pediatric Cardiopulmonary Resuscitation: Randomized Controlled Trial. J Med Internet Res. 2020 May 27;22(5):e17792. doi: 10.2196/17792. PMID 32292179
- [Background] Corazza F, Arpone M, Tardini G, Stritoni V, Mormando G, Graziano A, Navalesi P, Fiorese E, Portalone S, De Luca M, Binotti M, Tortorolo L, Salvadei S, Nucci A, Monzani A, Genoni G, Bazo M, Cheng A, Frigo AC, Da Dalt L, Bressan S. Effectiveness of a Novel Tablet Application in Reducing Guideline Deviations During Pediatric Cardiac Arrest: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2327272. doi: 10.1001/jamanetworkopen.2023.27272. PMID 37535352
- [Background] Corazza F, Stritoni V, Martinolli F, Daverio M, Binotti M, Genoni G, Ingrassia PL, De Luca M, Palmas G, Maccora I, Frigo AC, Da Dalt L, Bressan S. Adherence to guideline recommendations in the management of pediatric cardiac arrest: a multicentre observational simulation-based study. Eur J Emerg Med. 2022 Aug 1;29(4):271-278. doi: 10.1097/MEJ.0000000000000923. Epub 2022 Mar 29. PMID 35404331
- [Background] Corazza F, Snijders D, Arpone M, Stritoni V, Martinolli F, Daverio M, Losi MG, Soldi L, Tesauri F, Da Dalt L, Bressan S. Development and Usability of a Novel Interactive Tablet App (PediAppRREST) to Support the Management of Pediatric Cardiac Arrest: Pilot High-Fidelity Simulation-Based Study. JMIR Mhealth Uhealth. 2020 Oct 1;8(10):e19070. doi: 10.2196/19070. PMID 32788142
- [Background] Kruse CS, Krowski N, Rodriguez B, Tran L, Vela J, Brooks M. Telehealth and patient satisfaction: a systematic review and narrative analysis. BMJ Open. 2017 Aug 3;7(8):e016242. doi: 10.1136/bmjopen-2017-016242. PMID 28775188
- [Background] Cooper S, Cant R, Porter J, Sellick K, Somers G, Kinsman L, Nestel D. Rating medical emergency teamwork performance: development of the Team Emergency Assessment Measure (TEAM). Resuscitation. 2010 Apr;81(4):446-52. doi: 10.1016/j.resuscitation.2009.11.027. Epub 2010 Feb 1. PMID 20117874